CLINICAL TRIAL: NCT00244868
Title: Facilitating Decision Making in Advanced Cancer Patients
Brief Title: Computer-Based Survey and Communication Aid in Improving Physician-Patient Communication and Treatment Decision Making in Patients With Metastatic Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fox Chase Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized
Other Study IDs: CDR0000442928; FCCC-03826; FCCC-NCI-FC03CC9; NU-119-385
Record Dates: First submitted 2005-10-25; First posted 2005-10-27 (Estimated); Last update posted 2013-01-29 (Estimated); Status verified 2013-01

CONDITIONS: Metastatic Cancer; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific; metastatic cancer
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Counseling; Early Intervention, Educational

INTERVENTIONS:
Other: counseling intervention
Other: educational intervention

SUMMARY:
RATIONALE: A computer-based survey and communication aid may help physicians and patients to communicate better and help make treatment decisions easier.

PURPOSE: This phase III randomized clinical trial is studying how well giving a computer-based survey together with a communication aid works compared to a computer-based survey alone in improving physician-patient communication and treatment decision making in patients with metastatic cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare satisfaction with physician-patient communication and decisional conflict in patients with metastatic cancer undergoing a computer-based survey with vs without a communication aid.
* Compare patient expectations regarding potential benefits and adverse reactions associated with treatment options in patients undergoing the computer-based survey and communication aid.
* Compare the content of physician-patient consultations in patients undergoing the computer-based survey and communication aid.

OUTLINE: This is a randomized, controlled, multicenter study.

Patients are randomized to 1 of 3 study arms.

* Arm I (generic computer-based survey): Patients complete a 45- to 60-minute generic computer-based survey that assesses demographics, familiarity and comfort with computers, treatment history, and affective elements.
* Arm II (targeted computer-based survey and communication aid with physician summary report): Patients complete a 45- to 60-minute targeted computer-based survey assessing patient values, information needs, and distress. Patients then complete a targeted computer-based communication aid that addresses cognitive and affective components of cancer treatment education and provides communication skills training. After completion of the survey and communication aid, a summary report of the survey results is generated and provided to the patient's physician.
* Arm III (targeted computer-based survey and communication aid): Patients complete a targeted computer-based survey and communication aid as in arm II. No summary report is provided to the physician.

After completion of a computer-based survey and communication aid, all patients undergo a consultation with their physician. A randomized subset of 25% of physician consultations* are audiotaped and later analyzed. Patients complete a 15-minute written survey after completion of the physician consultation and then at 3 months.

NOTE: *Patients are stratified according to study arm (I vs II vs III) and consulting physician gender for this randomization.

PROJECTED ACCRUAL: A total of 720 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Documented metastatic malignancy
* First visit with medical oncologist at study site

PATIENT CHARACTERISTICS:

Performance status

* Not specified

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* Not specified

Renal

* Not specified

Other

* Able to read and speak English

PRIOR CONCURRENT THERAPY: Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 720 (Estimated)
Dates: Start 2003-07; Primary Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Satisfaction with patient-physician communication by Medical Interview Satisfaction Survey and Face Valid Survey given immediately after the first consultation
Assess decisional conflict by Decisional Conflict Scale immediately after the first consultation and at 3 months after study completion
Expectations regarding potential benefits and adverse reactions associated with treatment options by Treatment Options Expectations Scale given immediately after the first consultation and at 3 months after study completion
Assess content of consultation by applying a coding scheme to transcripts and design yes/no questions immediately after the first consultation

CONTACTS AND LOCATIONS:
Overall Officials: Neal J. Meropol, MD, Principal Investigator — Fox Chase Cancer Center
Locations (3):
- United States (3):
  - Robert H. Lurie Comprehensive Cancer Center at Northwestern University, Chicago, Illinois
  - Fox Chase Cancer Center - Philadelphia, Philadelphia, Pennsylvania
  - MBCCOP - Meharry Medical College - Nashville, Nashville, Tennessee

REFERENCES:
- [Result] Meropol NJ, Egleston BL, Buzaglo JS, Benson AB 3rd, Cegala DJ, Diefenbach MA, Fleisher L, Miller SM, Sulmasy DP, Weinfurt KP; CONNECT Study Research Group. Cancer patient preferences for quality and length of life. Cancer. 2008 Dec 15;113(12):3459-66. doi: 10.1002/cncr.23968. PMID 18988231